CLINICAL TRIAL: NCT02964117
Title: Associations Between Air Pollutants Exposures and Respiratory System Study
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Collaborators: Peking University (Other)
Responsible Party: Principal Investigator, Bei He, Clinical Professor, Peking University Third Hospital
Other Study IDs: Apers Study
Record Dates: First submitted 2016-10-31; First posted 2016-11-15 (Estimated); Last update posted 2016-11-15 (Estimated); Status verified 2016-11

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: Chronic Obstructive Pulmonary Disease
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine,Blood,Sputum and Exhaled breath condensate
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Epidemiological investigations has suggested exposure to air pollution linked with respiratory disease, especially chronic obstructive pulmonary disease. However, the potential mechanisms of adverse effects remains scare. The present study will assess the association between air pollutants and respiratory related parameters to elucidate possible mechanisms.

ELIGIBILITY:
Inclusion Criteria:

* Long-term residents, aged >23 and <82 years

Exclusion Criteria:

* Severe cardiopulmonary diseases, active inflammatory diseases, cancer

Ages: 23 Years to 82 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects including health volunteers and COPD patients,both of them without severe cardiopulmonary diseases and long-term residents in Beijing
Sampling Method: Non-Probability Sample
Enrollment: 106 (Actual)
Dates: Start 2014-11; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Lung Function indices were performed in peking university third hospital | Repeated-measure study was conducted from November,2014 to January,2016,lung function was measured by every four months
  Lung Function indices including FEV1(ml), FVC(ml),the ratio of FEV1/FVC et, al.. When we perform data analysis,these parameters will be expressed as the percentage of the predicted values based on the subject-specific sex, age,height and weight.

SECONDARY OUTCOMES:
Inflammation related biomarkers were measured by flow cytometry | Repeated-measure study was conducted from November,2014 to January,2016,biomarkers were measured by every four months
  Inflammation related factors including IL,TNFa et, al. all biomarkers units are pg/ml.

CONTACTS AND LOCATIONS:
Overall Officials: Bei He, MD/Ph.D, Study Director — Peking University Third Hospital